CLINICAL TRIAL: NCT01316861
Title: A Prospective, Randomized, Multicenter Study of the Efficacy and Safety of Oral Acarbose Treatment in Patients With Type 2 Diabetes Mellitus
Brief Title: Efficacy and Safety of Oral Acarbose Treatment in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EMSAGL0110
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2013-09-25 (Estimated); Status verified 2013-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EMS Acarbose (Experimental)
  Interventions: Drug: EMS Acarbose
- Bayer Acarbose (Active Comparator)
  Interventions: Drug: Bayer Acarbose

INTERVENTIONS:
Drug: EMS Acarbose — EMS Acarbose 50 mg 3 times a day
  Arms: EMS Acarbose
Drug: Bayer Acarbose — Bayer Acarbose 50 mg 3 times a day
  Arms: Bayer Acarbose

SUMMARY:
The Purpose of This Study is to Evaluate the Efficacy and Safety of Acarbose in Type 2 Diabetic Patients Using Two Different Formulations of Acarbose 50mg.

DETAILED DESCRIPTION:
Study Design:

* Multicenter
* Phase III
* Randomized
* Double Blind
* Prospective and Comparative
* Experiment duration: 105 days
* 5 visits
* Efficacy
* Adverse event

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to understand the study procedures agree to participate and give written consent.
* Diagnosed with type 2 diabetes mellitus (t2dm)b
* Female patients of childbearing potential (i.e., ovulating, pre-menopausal, not surgically sterile) which agree to use a medically accepted contraceptive regimen for the duration of the study.

Exclusion Criteria:

* Pregnancy or risk of pregnancy.
* Lactation
* Any pathology or past medical condition that can interfere with this protocol
* Other conditions deemed reasonable by the medical investigator as to the disqualification of the individual from study participation.
* Known hypersensitivity / intolerance to acarbose or any of its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2012-09; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Glycosylated hemoglobin (HbA1c) | Change from baseline to day 98

SECONDARY OUTCOMES:
Decrease in mean Fasting Plasma Glucose (FPG) | Change from baseline to day 14, 28, 42, 70 and 98
Safety will be evaluated by the Adverse events occurence | Day 105
  Adverse events will be collected and followed in order to evaluate safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Pinho, MD, Study Director — EMS S/A
Locations (1):
- Marcio Antonio Pereira Clinica, São José dos Campos, São Paulo, Brazil